CLINICAL TRIAL: NCT01197547
Title: Genesys HTA Post Approval Registry A Multi-center, Single-arm, Prospective Registry of the Genesys HTA System for the Treatment of Menorrhagia
Brief Title: Registry Study of Genesys HTA for Treatment of Menorrhagia
Acronym: Genesys HTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minerva Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U8088
Record Dates: First submitted 2010-09-01; First posted 2010-09-09 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2017-04

CONDITIONS: Menorrhagia
Keywords: Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genesys HTA (Other): Genesys HTA Endometrial Ablation
  Interventions: Device: Genesys HTA

INTERVENTIONS:
Device: Genesys HTA — Genesys HTA Endometrial Ablation
  Other Names: Genesys HTA Endometrial Ablation

SUMMARY:
This is a clinical registry of an FDA approved device system called the Genesys Hydro ThermAblatorTM (HTA) system (Boston Scientific). The HTA system's intended use is to be inserted, by a trained physician, into the uterus, where it will fill and circulate fluid that is warm enough to change the characteristics of the uterine lining. This is done with the anticipated result of improving menstrual bleeding symptoms.

The purpose of this FDA-mandated registry is to obtain clinical experience on the use the Genesys HTA™ system, under normal clinical conditions, and document its safety and technical reliability.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet the approved indication for use to be considered for this registry.

Exclusion Criteria:

* All subjects contraindicated for the treatment of the Genesys HTA System per the Directions for Use will be excluded:

  1. The subject is pregnant or wants to be pregnant in the future
  2. The subject has known or suspected endometrial carcinoma or premalignant change of the endometrium, such as adenomatous hyperplasia
  3. The subject has active pelvic inflammatory disease or pyosalpinx
  4. The subject has hydrosalpinx
  5. The subject in whom a tight cervical seal cannot be established and maintained around the procedure sheath
  6. The subject has an anatomical condition (e.g. history of previous classical cesarean section or transmural myomectomy) or pathologic condition (e.g. long term medical therapy) that could lead to weakening of the myometrium
  7. The subject has an intrauterine device in place
  8. The subject has an active genital or urinary tract infection (e.g. cervicitis, endometritis, vaginitis, cystitis, etc.) at the time of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1014 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bowman, M.D., Study Director — Boston Scientific Corporation
Locations (19):
- United States (19):
  - Sharp Mary Birch, San Diego, California
  - Christiana Hospital, Newark, Delaware
  - Shelnutt Obstetrics and Gynecology, Athens, Georgia
  - Health South Surgecenter of Louisville, Louisville, Kentucky
  - Wayne State University Physician Group, Southfield, Michigan
  - Seven Hills OB GYN Associates, Cincinnati, Ohio
  - Complete Healthcare for Women, Columbus, Ohio
  - Associates in Women's Healthcare, Philadelphia, Pennsylvania
  - Schuykill Medical Center South, Pottsville, Pennsylvania
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - State of Franklin Healthcare Associates, Johnson City, Tennessee
  - Associates in Obstetrics and Gynecology, Bedford, Texas
  - Central Womens Care PA, Dallas, Texas
  - Doreen Moser, DO, Grapevine, Texas
  - MacArthur OBGYN, Irving, Texas
  - Personalized Women's Healthcare, Plano, Texas
  - Ogden Clinic, Ogden, Utah
  - Old Farm Obstetrics and Gynecology, Salt Lake City, Utah
  - Milwaukee ObGyn, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Genesys HTA
Started | 1014
Completed | 992 (992 Intent-To-Treat (ITT) 931 evaluable subjects)
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Genesys HTA
Number analyzed (Participants) | 1014
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1013
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1014
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1014

OUTCOME MEASURES:

1. Primary Outcome: Burn Rate
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Genesys HTA
Number analyzed (Participants) | 992
participants | 4

2. Secondary Outcome: Technical Malfunctions
Description: A secondary endpoint of the Genesys HTA Post Approval Study is to assess technical complaints (i.e. disposable and hardware issues). Technical complaints are issues related to system components encountered during the procedure such as error messages, problems with the connection, power, early incomplete procedure terminations, or display/user interface, or damage to the unit.
Time Frame: Day 1
Population: 992 patients = ITT population
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Genesys HTA
Number analyzed (Participants) | 992
percent of participants
  complaint - procedure stopped to prevent injury | .6 [.2 to 1.3]
  Subjects with At Least One Technical Complaint | 4.4 [3.2 to 5.9]
  Subjects with One Technical Complaint | 3.5 [2.5 to 4.9]
  Subjects with Two Technical Complaints | .9 [.4 to 1.7]
  Subjects with Three Technical Complaints | 0.0 [0.0 to 0.4]
  Subjects with More Than Three Technical Complaints | 0.0 [0.0 to 0.4]
  Subjects with 1+ Component with Tech Comp | 4.4 [3.2 to 5.9]
  Subjects with One Component with Technical Complai | 4.2 [3.1 to 5.7]
  Subjects with Two Component with Technical Complai | .2 [0.0 to 0.7]

3. Secondary Outcome: Serious Adverse Device Effect (SADE)
Description: A secondary endpoint of the Genesys HTA Post Approval Study is to assess Serious Adverse Device Effects. Per the approved protocol, an SADE is an adverse device effect resulting in any of the consequences characteristic of a serious adverse event, or that might have led to any of these consequences if suitable action had not been taken or intervention had not been made, or if circumstances had been less opportune.
Time Frame: Day 1
Population: 992 - Intent-To-Treat (ITT) population
Measure: Number; unit: number of participants
Units Other Than Participants: participants
Arm/Group | Genesys HTA
Number analyzed (Participants) | 992
number of participants
  Subjects with at least one Serious adverse event | 1
  Injury, poisoning and procedural complications | 1
  Thermal burn | 1

ADVERSE EVENTS:
Arm/Group | Genesys HTA
Serious Adverse Events (participants affected / at risk) | 1/992
Other Adverse Events (participants affected / at risk) | 3/992
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genesys HTA (N=992)
Burn (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than .3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genesys HTA (N=992)
Clinically Non-Significant Burn (Reproductive system and breast disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No